CLINICAL TRIAL: NCT06797323
Title: Evaluating the Feasibility of a Web-App for Pelvic Floor Health in Pregnant Women in the Ferrol Health Area: the WaPRUIN Study
Acronym: WaPRUIN
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad de Oviedo (Other)
Responsible Party: Principal Investigator, Raquel Iglesias Méndez, PhD candidate, Universidad de Oviedo
Other Study IDs: 2023/291
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy; Pelvic Floor Disorder
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women
  Interventions: Behavioral: Web-Based Application for Pelvic Floor Health

INTERVENTIONS:
Behavioral: Web-Based Application for Pelvic Floor Health — A user-friendly web application designed to provide educational resources, exercises, and interactive tools aimed at improving pelvic floor health in pregnant women.

SUMMARY:
This study aims to evaluate the feasibility of using a web-based application to improve pelvic floor health in pregnant women within the Ferrol Health Area, Spain. The intervention involves providing educational resources through a user-friendly digital platform, designed to empower women with knowledge about pelvic floor function and techniques for strengthening it during pregnancy.

The study hypothesizes that a web-based educational tool can effectively increase awareness, engagement, and adherence to pelvic floor exercises among pregnant women, thereby contributing to improved maternal health outcomes. Participants will include pregnant women from the Ferrol Health Area, who will voluntarily use the application during their pregnancy.

The study will assess outcomes related to usability, accessibility, and participant satisfaction with the application, as well as any improvements in pelvic floor-related health indicators. By addressing an important gap in maternal health education, this project has the potential to provide an innovative and scalable solution to enhance prenatal care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending their first prenatal consultation at the Hospital Arquitecto Marcide.
* Pregnant women who voluntarily consent to participate in the study by signing the informed consent form.

Exclusion Criteria:

* Pregnant women who do not have proficiency in the Spanish language.
* Limitations in using the web-app (e.g., physical, cognitive, or technological barriers).
* Lack of internet access.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of pregnant women from the Ferrol Health Area who receive prenatal care in the Gynecology and Obstetrics Department at Hospital Arquitecto Marcide.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Web-App Usage | From enrollment to the end of web application use at 8 weeks
  To evaluate the feasibility and usability of the "PelviEduca" web-app, which is designed to improve knowledge about pelvic floor health and related conditions during pregnancy in pregnant women within the Ferrol Health Area.

SECONDARY OUTCOMES:
Frequency of Web-App Use | From enrollment to the end of web application use at 8 weeks
  To analyze the frequency of use of the web-app by the participants during the study.
Relationship Between Usability and Participant Characteristics | From enrollment to the end of web application use at 8 weeks
  To describe the relationship between the feasibility and usability of the web-app and the personal characteristics of the participants.
Knowledge Improvement on Pelvic Floor Health | From enrollment to the end of web application use at 8 weeks
  To evaluate whether the use of the web-app contributes to an increase in knowledge regarding pelvic floor health during pregnancy among participants.
Effectiveness in Encouraging Pelvic Floor Exercises | From enrollment to the end of web application use at 8 weeks
  To determine the effectiveness of the web-app in promoting the practice of pelvic floor exercises among participants.
Prevalence of Urinary Incontinence at Inclusion | At baseline (time of enrollment)
  To describe the percentage of pregnant women presenting urinary incontinence at the time of enrolment in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Arquitecto Marcide Hospital, Ferrol, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The decision on whether to share individual participant data (IPD) will be made after the completion of the study and analysis of results. Further updates will be provided when available.